CLINICAL TRIAL: NCT06331936
Title: Improving Emotional Regulation Skills of Children in Difficulty in Shenzhen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: International Social Service Hong Kong Branch (Unknown)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Shenzhen Project
Record Dates: First submitted 2024-02-02; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Emotion Regulation; Parent-Child Relations; Happiness; Positive Affect
Keywords: children in need; teenagers from low socioeconomic family; randomized wait-list control trial
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Children will be randomly assigned to two groups: intervention and waitlist control groups. Children in the waitlist control group will receive experimental intervention after treatment for the experimental group finishes.
Who Masked: Participant
Masking Description: At the recruitment phase, the participants and the social workers who lead the intervention will not know which arm the participants will be assigned. A cluster of approximately 10 participants formed a group based on their attendance date in the intervention program. This group will be randomly assigned to one of the two intervention arms through pre-prepared randomization list calculated by random allocation software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm aims at improving children's emotional regulation skills.
  Interventions: Behavioral: Emotion regulation
- Control Arm (No Intervention): The control arm participants will not receive any interventions.

INTERVENTIONS:
Behavioral: Emotion regulation — Each participant will attend four intervention sessions. They will also be invited to a booster Session, where they will be invited for interviews to share what they have gained from the sessions. The contents of the intervention and the booster session are as follows: (1) understand emotions, (2) attention and positivity, (3) emotional regulation, (4) connectedness and intimacy, and (5) review and sharing.
  Arms: Intervention arm

SUMMARY:
The study aims to 1) improve the emotional regulation strategies of children in difficulty in Shenzhen, and 2) develop and publish a set of evidence-based intervention manuals for professional use. Based on the intervention manual design of the researchers' previous study conducted in Hong Kong, the current research revised the intervention manual to adapt to the context of mainland China. This study adopts a randomized wait-list control trial design. The researchers aim to recruit 200 children in difficulty aged 8 to 14 as participants and randomly assign them to an experimental and a wait-list control group with a ratio of 3:2. Each participant will attend four sessions of intervention and one booster session, and each session requires around 1.5 to 2 hours to complete. The participants will complete assessments before the first session of the intervention (T1), immediately after the fourth session of the intervention (T2), and one month after the completion of the intervention (T3). A qualitative assessment will also be conducted after the booster session.

DETAILED DESCRIPTION:
1. Context of study

   The target population of this study is children in difficulty, which is defined as children who come from one of the following three groups: (1) single-parent families, (2) low-income families, and (3) left-behind children. Children in difficulty are constantly exposed to multiple sources of stress, including parental psychological neglect, unstable family life, limited school-based social activities, and stereotypes. These factors can bring emotional fluctuations in children. If they are not handled properly, it may lead to bullying, family conflicts, and even suicide.
2. Target of emotional regulation

   There are still challenges and deficiencies in the coverage, quality, and synergy of emotional assistance services for children in need. This study helps children acquire emotional concepts and management skills and offers an evidence-based intervention framework for service providers.
3. Cultural and contextual considerations in the intervention feature

   The current research revised the intervention manual, which was developed in the context of Hong Kong to adapt to mainland China.
4. Procedure

The researchers aim to recruit 200 children in difficulty to participate in the study. The age range of the participants is between 8 and 14. The participants will be randomly assigned to an experimental or wait-list control group with a 3:2 ratio. Each participant will attend four intervention sessions. Each session requires around 1.5 to 2 hours to complete. The pre-test, post-test, and follow-up survey each requires around 30 minutes to complete. The surveys are conducted to assess the effectiveness of the emotional management intervention on children's emotional management skills and its correlation with mental health and family functioning among the participants.

ELIGIBILITY:
Inclusion Criteria:

* single-parent families
* low-income families
* left-behind children

Exclusion Criteria:

* a history of severe psychotic symptoms
* have previously participated in a similar intervention program

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
10-item Emotional Management Strategy Questionnaire | Baseline, week 4, week 8
  Emotional management strategy questionnaire is a 10-item scale assessing parents' and children's emotional management strategy. Possible scores for each item range from 1 (not at all) to 6 (everyday). Higher scores indicate more frequent use of emotional management strategy.
10-item Positive and Negative Affect Schedule | Baseline, week 4, week 8
  Positive and negative affect schedule is a 10-item scale assessing parents' and children's positive and negative affect. Possible scores for each item range from 1 (not at all) to 6 (everyday). Higher scores indicate more positive or negative affect.
Patient Health Questionnaire-9 | Baseline, week 4, week 8
  Patient health questionnaire assesses the depressive symptoms among parents and children. Possible scores for each item range from 1 (not at all) to 4 (everyday). Higher scores indicate more depressive symptoms.
Generalized Anxiety Disorder Scale | Baseline, week 4, week 8
  Generalized anxiety disorder questionnaire assesses the anxiety symptoms among parents and children. Possible scores for each item range from 1 (not at all) to 4 (everyday). Higher scores indicate more anxiety symptoms.
Subjective Happiness Scale | Baseline, week 4, week 8
  Subjective happiness scale is a 4-item scale assessing parents' and children's subjective happiness. Possible scores for each item range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate more subjective happiness.
Connor-Davidson Resilience Scale 10-Item | Baseline, week 4, week 8
  Connor-Davidson resilience scale assesses the individual resilience among parents and children. Possible scores for each item range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate greater resilience.
Child-Parent Relationship Scale | Baseline, week 4, week 8
  Child-parent relationship scale is a 4-item scale assessing the relationship between parents and children. Possible scores for each item range from 1 (very dissatisfied) to 6 (very satisfied). Higher scores indicate better satisfaction with parents.
Family Harmony Scale | Baseline, week 4, week 8
  Family harmony scale is an 8-item scale assessing the family harmony. Possible scores for each item range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate better family harmony.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy YU, Dr., Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data available to other researchers.

REFERENCES:
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Driscoll, K., & Pianta, R. C. (1992). Child-Parent Relationship Scale. Journal of Early Childhood and Infant Psychology. https://doi.org/10.1037/t16909-000
- [Background] Fabrizio CS, Lam TH, Hirschmann MR, Pang I, Yu NX, Wang X, Stewart SM. Parental emotional management benefits family relationships: A randomized controlled trial in Hong Kong, China. Behav Res Ther. 2015 Aug;71:115-24. doi: 10.1016/j.brat.2015.05.011. Epub 2015 Jun 4. PMID 26112397
- [Background] Kroenke, K., & Spitzer, R. L. (2002). The PHQ-9: A New Depression Diagnostic and Severity Measure. Psychiatric Annals, 32(9), 509-515. https://doi.org/10.3928/0048-5713-20020901-06
- [Background] Lyubomirsky, S., Lepper, H.S. A Measure of Subjective Happiness: Preliminary Reliability and Construct Validation. Social Indicators Research, 46, 137-155 (1999). https://doi.org/10.1023/A:1006824100041
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Yu, N. X., Kam-fung Liu, I., & Bu, H. (2021). Enhancing resilience in cross boundary families: A parent-child parallel group intervention. Journal of Social Work, 21(4), 651-675. https://doi.org/10.1177/1468017320919103
- [Background] Yu X, Tam WW, Wong PT, Lam TH, Stewart SM. The Patient Health Questionnaire-9 for measuring depressive symptoms among the general population in Hong Kong. Compr Psychiatry. 2012 Jan;53(1):95-102. doi: 10.1016/j.comppsych.2010.11.002. Epub 2010 Dec 28. PMID 21193179
- [Background] Zhang C, Wang T, Zeng P, Zhao M, Zhang G, Zhai S, Meng L, Wang Y, Liu D. Reliability, Validity, and Measurement Invariance of the General Anxiety Disorder Scale Among Chinese Medical University Students. Front Psychiatry. 2021 May 19;12:648755. doi: 10.3389/fpsyt.2021.648755. eCollection 2021. PMID 34093269